CLINICAL TRIAL: NCT00425919
Title: A 24-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Of The Safety And Efficacy Of PPM-204 In Subjects With Type 2 Diabetes
Brief Title: Study Evaluating PPM-204 In Subjects With Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated as a result of interim analysis not meeting predetermined criteria.
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3180A1-200
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: PPM-204

SUMMARY:
The purpose of this study is to learn whether PPM-204 has an effect on lowering blood glucose (blood sugar) levels and is safe in treating people with type 2 diabetes.

DETAILED DESCRIPTION:
The objectives of the study are to identify doses of PPM-204 that are therapeutically effective and well tolerated in improving glycemic control over 24 weeks of treatment in subjects with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-childbearing potential, 18 to 70 years old
* Subjects currently treated with diet and exercise alone and subjects receiving a single oral antidiabetic medication
* BMI > 23 and < 43
* For subjects currently treated with 1 antidiabetic medication: HbA1c is greater than or equal to 6.8% and less than or equal to 8.5%.
* For subjects not currently treated with antidiabetic medications: HbA1c is greater than or equal to 7.2% and less than or equal to 9.0%

Exclusion Criteria:

* Subjects requiring insulin therapy
* Subjects currently receiving 2 or more oral antidiabetic medications
* Subjects requiring systemic corticosteroids, unless treatment was discontinued at least 4 weeks before the screening visit
* Subjects receiving warfarin
* Subjects currently receiving thiazolidinediones, unless treatment was discontinued 8 weeks before the screening visit
* Significant diabetic complications (retinopathy, nephropathy, symptomatic neuropathy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose

SECONDARY OUTCOMES:
Mean changes of HbA1c, Fasting Insulin, HOMA-IR and QUICKI indices, Body weight, waist measurements, total cholesterol, LDL-C, HDL-C, total/HDL, apolipoprotein A-1 & B, triglycerides, free fatty acids, hs C-reactive protein, adiponectin, edema.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Argentina, Scheima@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com; Trial Manager, Principal Investigator — For Chile, scheima@wyeth.com; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Croatia, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For Hong Kong, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezzlj@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Russia, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Serbia, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For UK/Great Britian, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Ukraine, WVPIMED@wyeth.com
Locations (60):
- United States (11):
  - Artesia, California
  - Los Angeles, California
  - Chipley, Florida
  - Destin, Florida
  - Marianna, Florida
  - West Palm Beach, Florida
  - Omaha, Nebraska
  - New York, New York
  - Austin, Texas
  - Richmond, Virginia
  - Tacoma, Washington
- Argentina (5):
  - Buenos Aires
  - Corrientes
  - La Plata
  - Mar Del Plata Pcia de Bs. As
  - Ramos Mejia, Pcia de Bs.
- Australia (3):
  - Daws Park, South Australia
  - Keswick, South Australia
  - Box Hill, Victoria
- Vila Clementino - Sao Paulo, Brazil
- Canada (5):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Charlottetown, Prince Edward Island
  - Laval, Quebec
  - Saint-Janvier, Quebec
- Beijing, China
- Croatia (3):
  - Krapinske Toplice
  - Rijeka
  - Zagreb
- Greece (2):
  - Athens
  - Thessaloniki
- Wan Chai, Hong Kong
- India (5):
  - Bangalore, Karnataka
  - Kochi, Kerala
  - Pune, Maharashtra
  - Chennai, Tamil Nadu
  - Vellore, Tamil Nadu
- Italy (2):
  - Catanzaro
  - Pisa
- Mexico (5):
  - Aguascalientes
  - Mexico City
  - Miguel Hidalgo
  - Monterrey N.L
  - Tlapan
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (2):
  - Moscow
  - Saint Petersburg
- Belgrade, Serbia and Montenegro
- South Africa (4):
  - Port Elizabeth, Eastern Cape
  - Benoni, Gauteng
  - Pretoria, Gauteng
  - Temba, North West
- Ukraine (4):
  - Kharkiv
  - Kyiv
  - Poltava
  - Uzhhorod
- United Kingdom (3):
  - Dundee
  - Edinburgh
  - Livingston